CLINICAL TRIAL: NCT07033078
Title: Exploring Sleep, Mood, and Quality of Life Issues in Adolescents and Adults With Autism and Asperger
Brief Title: Sleep, Mood, and Quality of Life Issues in ASD Adolescents and Adults.
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400427B0
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Asperger Disorder; High Functioning Autism; Sleep; Polysomnography; Actigraphy
MeSH Terms: conditions — Autism Spectrum Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ASD
- Asperger

SUMMARY:
Autism Spectrum Disorder (ASD) presents unique challenges, particularly in sleep, mood, and quality of life for adolescents and adults. Due to the pressures of life they face, these groups may experience more severe sleep problems and emotional issue and associated issues than children. Current research on these sleep and emotional issues in older ASD individuals is limited, and there is a need for studies on various sleep and emotional problems they encounter. This study aims to compare sleep patterns in adolescents and adults with Asperger's syndrome and high-functioning autism using both subjective and objective measures, such as questionnaires and polysomnography. It also examines the factors influencing sleep, including cognitive function, emotional and behavioral problems, and quality of life. Additionally, the study evaluates the reliability and validity of the Chinese Social Responsiveness Scale-Adult Version in Taiwan. The expected outcome is that sleep and emotional issues in these populations are linked to anxiety, depression, poorer functioning, and lower quality of life.

DETAILED DESCRIPTION:
A.Background Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by core symptoms such as social communication difficulties and repetitive behaviors. Considering the challenges of employment and social environments for adult and adolescents with ASD, sleep problems, quality of life, and functioning may be more severely impacted in adults and adolescents than in children. However, there is few research on sleep problems in adult and adolescents with ASD, as well as a lack of studies on different types of sleep problems in adults and adolescents with ASD. Furthermore, the Social Responsiveness Scale (SRS) is a commonly used assessment tool for ASD, but there are currently lack of validation studies for the adult version of the scale in Taiwan, necessitating further exploration.

B.Purpose This study aims to compare sleep patterns in adults and adolescents with Asperger's syndrome and high-functioning autism using subjective and objective measures such as questionnaires, actigraphy, and PSG. We also explore these factors affecting sleep and related issues including cognitive function, emotional and behavioral problems, autism symptoms, and quality of life. This research will enhance our understanding of sleep problems in Asperger's syndrome and high-functioning autism, tracking the changes in sleep patterns of autism patients at different developmental stages, the relevance to quality of life and prognosis, and also evaluate the reliability and validity of the Chinese Social Responsiveness Scale-Adult Version.

C.Study design This study is a cross-sectional study consisting of two parts. The first part is a retrospective study that includes adolescents and adults with Asperger's syndrome and high-functioning autism who underwent overnight polysomnography in the past. Their sleep studies results and questionnaires were collected. The second part is a prospective study involving outpatient adolescents and adults with Asperger's syndrome and high-functioning autism who have not undergone polysomnography. After enrollment, they undergo sleep studies using subjective and objective measurements including the Pittsburgh Sleep Quality Index (PSQI), actigraphy, and polysomnography. They also complete questionnaires such as the Child Behavior Checklist (CBCL) for assessing emotional and behavioral problems, the Social Responsiveness Scale (SRS), the Aberrant Behavior Checklist (ABC), the Chinese version of the Swanson, Nolan, and Pelham IV Scale (SNAP-IV), and the Adult ADHD Self-Report Scale (ASRS) for assessing autism-related symptoms. Additionally, anxiety and depression symptoms are assessed using the Beck Anxiety Inventory (BAI) and the Beck Depression Inventory (BDI), respectively. The SF-36 Health Survey is used to evaluate quality of life. Correlation analyses are conducted, and comparisons are made with a control group of typically developing adults and adolescents.

D.Predicted results This study aim to predict that sleep patterns in adolescents and adults with autism are associated with depression, anxiety, poorer functioning, lower quality of life, autism symptoms, and poorer prognosis. Considering the increased stress of work and workplace adaptation difficulties in adults and adolescents, they are expected to experience more sleep problems compared to typically developing adults. Additionally, adults and adolescents with Asperger's syndrome and high-functioning autism are likely to exhibit different sleep patterns. Furthermore, additional analysis could be conducted on the reliability and validity of the Chinese version of the Social Responsiveness Scale for adults. The results could then be applied to adults with Autism Spectrum Disorder in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed by a psychiatrist as meeting the DSM-IV-TR diagnosis of Asperger's syndrome or autism.
2. Subjects were aged between 13-45 years old, male or female.
3. The subjects and their families agree to join the trial and sign the subject consent form.

Exclusion Criteria:

1. Cases where clinical assessment cannot be combined with sleep examination.
2. Cases where the intelligence test result showed that the full scale IQ was <70.
3. Those with serious physiological diseases, such as congenital heart disease, thyroid dysfunction, immune deficiency diseases, severe autoimmune diseases, brain injuries or severe organic brain diseases, which will affect the evaluation results.
4. Severe mental illness, such as severe schizophrenia, bipolar disorder, etc.
5. Not willing to participate in this study or unwilling to fill out the consent form.
6. Those who are not suitable to enter the trial after being evaluated by the PI and co-PI.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by core symptoms such as social communication difficulties and repetitive behaviors.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Actigraphy | 7 days
  Using actigraphy to assess the differences in sleep patterns between individuals with Autism Spectrum Disorder (ASD) and typically developing controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan